CLINICAL TRIAL: NCT06081881
Title: Predictors for Chronic Thromboembolic Pulmonary Hypertension After Pulmonary Embolism Episode
Brief Title: Chronic Thromboembolic Pulmonary Hypertension After Pulmonary Embolism
Status: Recruiting | Type: Observational
Sponsor: Ester Ashraf Faried Beshay (Other)
Responsible Party: Sponsor-Investigator, Ester Ashraf Faried Beshay, Physician Resident, Assiut University
Organization: Assiut University (Other)
Other Study IDs: CTEPH after pulmonary embolism
Record Dates: First submitted 2023-09-25; First posted 2023-10-13 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: CTEPH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to detect the incidence of CTEPH patients.

Primary outcome To predict CETHP in symptomatic patients after pulmonary embolism episode.

Secondary outcome:

On Echocardiography revealed RV dysfunction which are peak TR Velocity , the RV/LV basal diameter ratio, flattening of the IVS, RV acceleration time and/or midsystolic notching, IVC diameter with decreased inspiratory collapse and RA area.

DETAILED DESCRIPTION:
Chronic thrombo embolic pulmonary hypertension(CTEPH)is a progressive pulmonary vascular disease characterized by chronic obstruction of major pulmonary arteries with flow-limiting organized thrombi. In the clinical classification of the 6thWorld Symposium on Pulmonary Hypertension, CTEPH/chronic thromboembolic pulmonary disease(CTED)are in group4, labeled as PH due to pulmonary artery obstruction. CTEPH should be considered in PE patients if:(1)they report symptoms that could be related to CTEPH or with frank right heart failure,(2)the CTPA used to diagnose acute PE shows signs indicative of CTEPH,(3)they have risk factors or predisposing conditions for CTEPH. Recurrent venous thromboembolism(VTE),post-thrombotic syndrome, bleeding ,and functional limitations as important outcome measures of acute PE treatment , Dyspnea ,anxiety, chest pain ,post-thrombotic panic syndrome, and depression that lead to persistent functional limitations and/or decreased quality of life have been labeled as post-PE syndrome(PPS),includes CTEPH. Early diagnosis of CTEPH is important ,as it is the only form of PH that is potentially curable , but also challenging because signs of right heart failure only become evident in advanced disease stages and earlier disease stages are characterized by non specific or even absence of symptoms. The diagnostic work up of suspected CTEPH ,starts with trans thoracic Doppler echocardiography, In addition to the peak tricuspid regurgitation velocity , the right ventricle/left ventricle basal diameter ratio, flattening of the interventricular septum, right ventricular acceleration time and/or mid systolic notching, inferior vena cava diameter with decreased inspiratory collapse and right atrial area are used echocardiographic signs to assess the probability of PH.

ELIGIBILITY:
Inclusion Criteria:

Any patient diagnosed as acute pulmonary embolism ,aged between 18-80 years old which Pulmonary Embolism Severity Index (PESI) class III-V or sPESI ≥1,

Exclusion Criteria:

Secondary causes for pulmonary hypertension Severe kidney injury(eGFR>30 mg/dl/1.7m2) Hepatic affection Contraindication to anti-coagulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients underwent pulmonary embolism episodes
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of CTEHP in symptomatic patients after pulmonary embolism episode. | 3 years
  Incidence of CTEHP in symptomatic patients after pulmonary embolism episode.

SECONDARY OUTCOMES:
Measure of RV dysfunction by Echocardiography | 3 years
  Measure of RV dysfunction by Echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Ester A Faried, Resident, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt